CLINICAL TRIAL: NCT02378402
Title: Exploring Myocardial Lipid and Creatine as Imaging Biomarkers for Patients of Heart Failure
Brief Title: Myocardial Lipid and Creatine of Heart Failure on MRS
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Gigin Lin, Staff Radiologist, Chang Gung Memorial Hospital
Other Study IDs: 102-2772A3
Record Dates: First submitted 2015-02-27; First posted 2015-03-04 (Estimated); Results first posted 2019-10-21 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Myocardial Lipid
Keywords: Creatine; heart failure; lipid; MRS; myocardium
MeSH Terms: conditions — Heart Failure | interventions — Protons; Magnetic Resonance Spectroscopy; Spectrum Analysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Unstable HF group: Patients with acute HF episode with hospitalization treatment within 12 months, currently LVEF<50%. Proton (1H-) magnetic resonance (MR) spectroscopy.
  Interventions: Other: Proton (1H-) magnetic resonance (MR) spectroscopy
- Stable HF group: Patients with acute HF episode with hospitalization treatment within 12 months, LVEF>=50%. Proton (1H-) magnetic resonance (MR) spectroscopy.
  Interventions: Other: Proton (1H-) magnetic resonance (MR) spectroscopy
- Control group: Age- and gender-matched healthy volunteers recruited as normal control group. Proton (1H-) magnetic resonance (MR) spectroscopy.
  Interventions: Other: Proton (1H-) magnetic resonance (MR) spectroscopy

INTERVENTIONS:
Other: Proton (1H-) magnetic resonance (MR) spectroscopy — PRESS localized 1D MRS sequence was used on a 3-T MR system. The lipid resonances will be analyzed using the LC-Model algorithm, and a Cramer-Rao lower bound (CRLB) threshold of 50% was used as quality control. Resonances of fatty acid (FA, lipid resonances δ 0.9, 1.3 and 1.6 ppm) and polyunsaturated fatty acid (PUFA, lipid resonance δ 2.1 and 2.3, 2.8, 5.3 ppm) will be evaluated on MRS, with ratios normalized with total TG value.

SUMMARY:
The objective of this 3-year project is to develop myocardial MRS, in particular lipid (triglyceride) and creatine resonances, as imaging biomarkers for patients with heart failure (HF). Investigators will elucidate how and, to what extent, lipid and creatine levels of the heart contribute to heart failure. The first year is a cross-sectional study. Investigators aim to compare the MRS of normal subjects and that of stable HF patients in recovery with normal or impaired ejection fraction (EF). Total 60 subjects will be enrolled, with 20 subjects in each group. In the 2nd and 3rd years, investigators plan a prospective longitudinal study of 40 subjects. Enrolled patients will be evaluated with cardiac MRS at three time points, i.e., disease onset, 6 months and one year after treatment, and will be followed up until the end of this project (1.5~3-year follow up). In total 120 MR scans will be performed in the 2nd and 3rd years. The resonances from cardiac MRS, including creatine and lipids, will be correlated with the disease course, patient biochemistry data and clinical outcome. Investigators expect to make MRS to become an integral part of a clinical cardiac MR protocol.

DETAILED DESCRIPTION:
Heart failure (HF) is a major societal burden due to its high prevalence, poor prognosis and high cost. A potential therapeutic target is to supply the energy-starved heart. Lipid content of the heart is highly dynamic and myocardial lipid overload has been implicated in the pathophysiology of cardiac disease. The measurement of total creatine, a crucial actor in the creatine kinase system, gives an insight into the energy storage and buffering capacity in the heart. Magnetic Resonance Spectroscopy (MRS) is an imaging technique that allows non-invasive biochemical analysis in the clinical setting using routine MR scanner. It has the combined advantages of inherently providing molecular information, being free of ionizing radiation, and not requiring administration of external tracers. The objective of this 3-year project is to develop myocardial MRS, in particular lipid (triglyceride) and creatine resonances, as imaging biomarkers for patients with heart failure (HF). Investigators will elucidate how and, to what extent, lipid and creatine levels of the heart contribute to heart failure. The first year is a cross-sectional study. Investigators aim to compare the MRS of normal subjects and that of stable HF patients in recovery with normal or impaired ejection fraction (EF). Total 60 subjects will be enrolled, with 20 subjects in each group. In the 2nd and 3rd years, investigators plan a prospective longitudinal study of 40 subjects. Enrolled patients will be evaluated with cardiac MRS at three time points, i.e., disease onset, 6 months and one year after treatment, and will be followed up until the end of this project (1.5~3-year follow up). In total 120 MR scans will be performed in the 2nd and 3rd years. The resonances from cardiac MRS, including creatine and lipids, will be correlated with the disease course, patient biochemistry data and clinical outcome. Investigators expect to make MRS to become an integral part of a clinical cardiac MR protocol. The advance in knowledge is to prove the association between heart failure and myocardial impairment in lipids and/or creatine. The knowledge gained from MRS could potentially translate as a non-invasive biomarker for heart failure patients. This biomarker can help to early detect treatable causes of HF, and to monitor and evaluate treatment response in a non-invasive fashion. The inherited non-invasiveness and non-radiation nature makes MR an ideal technique for clinical application and biotechnology development.

ELIGIBILITY:
Inclusion Criteria:

1. heart failure patients diagnosed in the Keelung Chang Gung Memorial Hospital
2. without previous history of coronary artery disease
3. patients must be ≥ 20 and ≤ 80 years of age
4. patients must be willing to undergo standard treatment and follow up in the Heart Failure Center
5. patients must be able to give informed consent.

Exclusion Criteria:

1. patients who are judged to be noncompliant to treatment or not accessible for follow up
2. patients with contraindications to MR scanning, such as claustrophobia, cardiac pacemaker, metal implants, or unable to cooperate for MRI study due to mental status
3. Severe renal function impairment (glomerular filtration rate less than 30 mL/min/1.73m2)
4. pregnant or breast-feeding status
5. history of open-heart surgery.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with acute HF episode with hospitalization treatment within 12 months were enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2014-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiology, Chang Gung Memorial Hospital, Guishan, Taoyuan, Taiwan

REFERENCES:
- [Background] Liao PA, Lin G, Tsai SY, Wang CH, Juan YH, Lin YC, Wu MT, Yang LY, Liu MH, Chang TC, Lin YC, Huang YC, Huang PC, Wang JJ, Ng SH, Ng KK. Myocardial triglyceride content at 3 T cardiovascular magnetic resonance and left ventricular systolic function: a cross-sectional study in patients hospitalized with acute heart failure. J Cardiovasc Magn Reson. 2016 Feb 5;18:9. doi: 10.1186/s12968-016-0228-3. PMID 26850626
- See also: Myocardial triglyceride content at 3 T cardiovascular magnetic resonance and left ventricular systolic function: a cross-sectional study in patients hospitalized with acute heart failure. — http://www.ncbi.nlm.nih.gov/pubmed/26850626
- Available data/document: Clinical Study Report: ClinicalTrials.gov/NCT02378402 — http://jcmr-online.biomedcentral.com/articles/10.1186/s12968-016-0228-3

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Unstable HF Group | Stable HF Group | Control Group
Started | 25 | 25 | 21
Completed | 25 | 23 | 21
Not Completed | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Unstable HF Group | Stable HF Group | Control Group | Total
Number analyzed (Participants) | 25 | 23 | 21 | 69
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 24 | 20 | 18 | 62
  >=65 years | 1 | 3 | 3 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.0 (7.7) | 56.1 (8.7) | 58.9 (7.2) | 56.9 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 4 | 9
  Male | 21 | 22 | 17 | 60

OUTCOME MEASURES:

1. Primary Outcome: Myocaridal Lipid on MRS
Description: We quantified the total myocardial TG resonance as well as its components including FA (lipid resonances δ 0.9, 1.3 and 1.6 ppm) and UFA (lipid resonance δ 2.1 and 2.3, 2.8, 5.3 ppm) from water-suppressed spectra. We also determined the water resonance (~ δ 4.7 ppm) from spectra without water suppression. Myocardial TG content relative to water as well as relative amounts of myocardial TG was calculated from the available data.
Time Frame: 12 month
Measure: Mean (Standard Deviation); unit: ratios
Groups:
- Unstable HF Group: Patients with acute HF episode with hospitalization treatment within 12 months, currently LVEF<50%. Proton (1H-) magnetic resonance (MR) spectroscopy.
  Proton (1H-) magnetic resonance (MR) spectroscopy: PRESS localized 1D MRS sequence was used on a 3-T MR system. The lipid resonances will be analyzed using the LC-Model algorithm, and a Cramer-Rao lower bound (CRLB) threshold of 50% was used as quality control. We quantified the total myocardial TG resonance as well as its components including FA (lipid resonances δ 0.9, 1.3 and 1.6 ppm) and UFA (lipid resonance δ 2.1 and 2.3, 2.8, 5.3 ppm) from water-suppressed spectra. We also determined the water resonance (~ δ 4.7 ppm) from spectra without water suppression. Myocardial TG content relative to water as well as relative amounts of myocardial TG was calculated from the available data.
- Stable HF Group: Patients with acute HF episode with hospitalization treatment within 12 months, LVEF>=50%. Proton (1H-) magnetic resonance (MR) spectroscopy.
  Proton (1H-) magnetic resonance (MR) spectroscopy: PRESS localized 1D MRS sequence was used on a 3-T MR system. The lipid resonances will be analyzed using the LC-Model algorithm, and a Cramer-Rao lower bound (CRLB) threshold of 50% was used as quality control. We quantified the total myocardial TG resonance as well as its components including FA (lipid resonances δ 0.9, 1.3 and 1.6 ppm) and UFA (lipid resonance δ 2.1 and 2.3, 2.8, 5.3 ppm) from water-suppressed spectra. We also determined the water resonance (~ δ 4.7 ppm) from spectra without water suppression. Myocardial TG content relative to water as well as relative amounts of myocardial TG was calculated from the available data.
- Control Group: Age- and gender-matched healthy volunteers recruited as normal control group. Proton (1H-) magnetic resonance (MR) spectroscopy.
  Proton (1H-) magnetic resonance (MR) spectroscopy: PRESS localized 1D MRS sequence was used on a 3-T MR system. The lipid resonances will be analyzed using the LC-Model algorithm, and a Cramer-Rao lower bound (CRLB) threshold of 50% was used as quality control. We quantified the total myocardial TG resonance as well as its components including FA (lipid resonances δ 0.9, 1.3 and 1.6 ppm) and UFA (lipid resonance δ 2.1 and 2.3, 2.8, 5.3 ppm) from water-suppressed spectra. We also determined the water resonance (~ δ 4.7 ppm) from spectra without water suppression. Myocardial TG content relative to water as well as relative amounts of myocardial TG was calculated from the available data.
Arm/Group | Unstable HF Group | Stable HF Group | Control Group
Number analyzed (Participants) | 25 | 23 | 21
ratios
  triglyceride/water | 1.72 (2.63) | 1.18 (1.82) | 1.53 (1.78)
  fatty acids/water | 0.93 (2.13) | 0.97 (1.64) | 1.39 (1.67)
  unsaturated fatty acids/water | 0.79 (1.38) | 0.21 (0.28) | 0.14 (0.20)
  fatty acids/triglyceride | 0.53 (0.41) | 0.68 (0.40) | 0.71 (0.32)
  unsaturated fatty acids/triglyceride | 0.47 (0.41) | 0.32 (0.40) | 0.29 (0.32)

ADVERSE EVENTS:
Time Frame: Patients will be clinically followed on a monthly basis by a dedicated HF team, up to 3 year.
Arm/Group | Unstable HF Group | Stable HF Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/23 | 0/21
Other Adverse Events (participants affected / at risk) | 0/25 | 0/23 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes